CLINICAL TRIAL: NCT04482400
Title: Reducing Sedentary Time Using an Innovative mHealth Intervention Among Total Knee Replacement Patients
Brief Title: Technology Interventions to Improve Outcomes After Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Northwestern University (Other); Prisma Health-Midlands (Other)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00092132
Record Dates: First submitted 2020-07-16; First posted 2020-07-22 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Knee Arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEAT!2 (Experimental): Participants randomized to this arm will use the NEAT!2 app and receive biweekly coaching calls for 8 weeks, and monthly maintenance calls between months 2-5.
  Interventions: Behavioral: NEAT!2
- MyKneeGuide (Active Comparator): Participants randomized to this arm will use the MyKneeGuide app/website and receive biweekly coaching calls for 8 weeks, and monthly maintenance calls between months 2-5.
  Interventions: Behavioral: MyKneeGuide

INTERVENTIONS:
Behavioral: NEAT!2 — 8 week sedentary reduction program
  Arms: NEAT!2
Behavioral: MyKneeGuide — 8 week surgery recovery education program
  Arms: MyKneeGuide

SUMMARY:
The purpose of this study is to examine the effects of two technology interventions on health outcomes (e.g., physical activity, sedentary behavior, physical function, pain) after knee replacement at 2 and 5 months .

DETAILED DESCRIPTION:
Two 8 week technology interventions will be examined and consist of the use of an app and/or website and regular calls. Assessments to examine outcomes will be completed at baseline, as well as at 2 and 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Be 40-79 years of age
* Had unilateral knee replacement within last 12 months
* Have an Android or iOS smartphone that is accessible and near them the majority of the day
* Be willing to download the study applications on their smartphone
* Spend at least 7 hours/day sitting
* Be English speaking

Exclusion Criteria:

* Have any contraindications to activity
* Have a mobility limiting comorbidity
* Have a scheduled surgery within the next 6 months
* Do not have ≥4 days of valid accelerometer (>=10 hours) wear at baseline.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Objectively Measured (Actigraph) Sedentary Behavior at 2 months | 2 months - baseline
  change sedentary behavior (<100 counts/minute) measured with Actigraph accelerometers between baseline and 3 months
Change in Objectively Measured (Actigraph) Sedentary Behavior at 5 months | 5 months - baseline
  change in sedentary behavior (<100 counts/minute) measured with Actigraph accelerometers between baseline and 6 months

SECONDARY OUTCOMES:
Change in Physical Function | 5 months after surgery
  Six minute walk test
Change in WOMAC Pain Subscale | 5 months after surgery
  WOMAC Pain Subscale - Scores range from 0 (no pain) to 20 (maximal pain)
Total physical activity measured by Actigraph accelerometers | 5 months after surgery
  objectively measured light, moderate and vigorous activity (>= 100 counts/min) by Actigraph accelerometers
Adherence to NEAT!2 calls | 2 months
  Number of calls completed
Adherence to NEAT!2 app | 2 months
  total days NEAT! app was used
Response to NEAT!2 prompts | 2 months
  percentage of notifications in which a transition from sitting to standing was detected
Change in physical function via chair stand test | 5 months after surgery
  Chair stand test

OTHER OUTCOMES:
Change in physical function via timed up and go | 5 months after surgery
  Timed up and go test
Change in Knee Symptoms - KOOS pain | 5 months
  KOOS pain subcale (0 indicates extreme problems, 100 no problems)
Change in Knee Symptoms - KOOS symptoms | 2 months
  KOOS symptoms subcale (0 indicates extreme problems, 100 no problems)
Change in Knee Symptoms - KOOS ADL | 5 months
  KOOS ADL subcale (0 indicates extreme problems, 100 no problems)
Change in Knee Symptoms - KOOS sport/rec | 5 months
  KOOS sport/rec subcale (0 indicates extreme problems, 100 no problems)
Change in Knee Symptoms - KOOS QoL | 5 months
  KOOS QOL subcales (0 indicates extreme problems, 100 no problems)
Change in knee symptoms via WOMAC | 5 months
  WOMAC total score (pain, stiffness, and function) - Scores range from 0 (no problems) to 96 (extreme problems)
Change in sedentary time via activPAL accelerometers | 5 months
  activPAL accelerometer
Patient Reported outcomes - Mobility - T-Score | 5 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) - T score of 50 represents average for general population (scores higher than 50 represent better function and mobility)
Patient Reported outcomes - global health - T-Score | 5 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health - T score of 50 represents average for general population (scores higher than 50 represent better health)
Patient Reported outcomes - sleep disturbance - T-Score | 5 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep disturbance - T score of 50 represents average for general population (scores higher than 50 represent worse sleep disturbance)
Change in habit strength | 5 months
  adapted self-report habit index
Change in sedentary time via SIT-Q | 5 months
  SIT-Q
Weight | 5 months
  Change in weight

CONTACTS AND LOCATIONS:
Overall Officials: Christine Pellegrini, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be made available 12 months after the primary manuscript is published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after primary manuscripts are published